CLINICAL TRIAL: NCT05728918
Title: Effectiveness of Antrodia Cinnamomea Mycelia on Improving Immune Response in Subhealth People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Greenyn Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-111-091
Record Dates: First submitted 2023-02-01; First posted 2023-02-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Fatigue Syndrome, Chronic; Cold
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placeo group
  Interventions: Dietary Supplement: Placebo
- Treatment (Experimental): Experimental group
  Interventions: Dietary Supplement: Antrodia cinnamomea mycelia

INTERVENTIONS:
Dietary Supplement: Antrodia cinnamomea mycelia — Antrodia cinnamomea mycelia capsule, two capsules/day (600 mg/day) for 3 months
  Arms: Treatment
Dietary Supplement: Placebo — Placebo capsule, two capsules/day (600 mg/day) for 3 months
  Arms: Placebo

SUMMARY:
This study aims to assess the effect of Antrodia cinnamomea mycelia on immune modulation in subhealth people.

DETAILED DESCRIPTION:
This study aims to assess the effect of Antrodia cinnamomea mycelia on immune modulation in subhealth people: a randomized, double-blind, placebo-controlled, and parallel clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are easy to feel fatigued
* Subjects have poor sleep quality

Exclusion Criteria:

* Pregnant women or preparing for pregnancy.
* Lactating women.
* Women gave birth 6 months before the study.
* Poor kindy and livers funcitons
* Severe cardiovascular or other chronic diseases
* Alcohol abuser
* Using immune-associated supplements

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Immune analysis | Baseline up to 4 weeks
  Changes in T cell markers of 29 participants will be analyzed between baseline and week 4.
Immune analysis | Baseline up to 4 weeks
  Changes in B cell markers of 29 participants will be analyzed between baseline and week 4.
Antibody analysis | Baseline up to 4 weeks
  Changes in IgA levels of 29 participants will be analyzed between baseline and week 4.
Antibody analysis | Baseline up to 4 weeks
  Changes in IgD levels of 29 participants will be analyzed between baseline and week 4.
Antibody analysis | Baseline up to 4 weeks
  Changes in IgG levels of 29 participants will be analyzed between baseline and week 4.
Antibody analysis | Baseline up to 4 weeks
  Changes in IgE levels of 29 participants will be analyzed between baseline and week 4.
Antibody analysis | Baseline up to 4 weeks
  Changes in IgM levels of 29 participants will be analyzed between baseline and week 4.
Cytokine analysis | Baseline up to 4 weeks
  Changes in IL-1beta levels of 29 participants will be analyzed between baseline and week 4.
Cytokine analysis | Baseline up to 4 weeks
  Changes in IL-4 levels of 29 participants will be analyzed between baseline and week 4.
Cytokine analysis | Baseline up to 4 weeks
  Changes in IL-6 levels of 29 participants will be analyzed between baseline and week 4.
Cytokine analysis | Baseline up to 4 weeks
  Changes inFN-gamma levels of 29 participants will be analyzed between baseline and week 4.
Cytokine analysis | Baseline up to 4 weeks
  Changes in TNF-alpha levels of 29 participants will be analyzed between baseline and week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shun Wu, MD, Principal Investigator — WanFang Hospital
Locations (1):
- WanFang Hospital, Taipei, Taiwan